CLINICAL TRIAL: NCT04104464
Title: Patient Reported Outcomes for Vascular Malformations EmbolizatioN (PROVEN)
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00205322
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Vascular Malformations; VM - Vascular Malformation
Keywords: vascular malformation; VM
MeSH Terms: conditions — Vascular Malformations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a standardized assessment for patients treated for venous malformations (VM).

Venous malformations result from the abnormal development of veins which may result in pain, swelling, bleeding, functional impairment, disfigurement, and psychological distress. The impact of VM on patient quality of life varies based on the location and size of the malformation.

A patient reported outcome (PRO) is a patient's own account of patient's health condition. PRO measures are valued to clinicians, as many treatment effects are known only to the patient. No studies to date have analyzed the validity of existing PRO measures for VM patients.

Current assessment does not include all symptoms or take in to account the relevance of VM location. Past studies show a discrepancy between treatment outcomes reported by patients and physicians. Therefore, there is a need to develop VM-specific PROs to better understand the effectiveness and benefits of treatment for VM.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female pediatric patients, aged between 0-17 with diagnosis of vascular malformations.
* Male and Female adult patients aged 18-100 with diagnosis of vascular malformations.
* Vascular malformation symptoms significant enough to seek treatment.

Exclusion Criteria:

* Patients with extensive VM not suitable for sclerotherapy.
* Prior therapy for treatment of a VM within 3 months.
* Condition or impairment that may render the patient unable to take part in the study (e.g. cognitive, sight, hearing, etc.).

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Vascular Malformation patients treated in the Interventional Radiology clinic.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported VM pain | 1 month, 3 months and 6 months post-procedure; and all subsequent visits up to 1 year
  Patients are asked to rate pain associated with VM during the past seven days on a 0-10 scale.
Change in patient reported VM impact on daily life | 1 month, 3 months and 6 months post-procedure; and all subsequent visits up to 1 year
  Patients are asked to rate the impact that their VM has on daily life with the options "Not at all", "A little bit", "Somewhat", "Quite a bit" or "Very Much".
Change in patient reported efficacy of treatment | 1 month, 3 months and 6 months post-procedure; and all subsequent visits up to 1 year
  Patients are asked to rate the efficacy of their treatment with the options "Not at all", "A little bit", "Somewhat", "Quite a bit" or "Very Much".
Change in patient reported relevancy of the PROVEN Questionnaire | 1 month, 3 months and 6 months post-procedure; and all subsequent visits up to 1 year
  Patients are asked to rate the personal relevancy and clarity of the survey questions with the options "Not at all", "A little bit", "Somewhat", "Quite a bit" or "Very Much".

CONTACTS AND LOCATIONS:
Overall Officials: Clifford R Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States